CLINICAL TRIAL: NCT07053592
Title: Enhancing Well-being Through Beauty: Applying Experiential Learning in Senior Beauty and Health Care Courses for Community Practice and Effectiveness Evaluation
Brief Title: Community Beauty and Health Program for Older Adults: An Experiential Learning Trial
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 202500403B0
Record Dates: First submitted 2025-07-07; First posted 2025-07-08 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Aged; Experiential Learning; Health Education
MeSH Terms: conditions — Health Education

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Learning Intervention Group (Experimental): Participants in this group will receive a curriculum intervention designed to improve attitudes and learning outcomes toward older adults. The course includes interactive teaching and adopts mixed research methods for effectiveness evaluation. Quantitative data were collected through pre- and post-test questionnaires to assess students' attitudes towards the elderly, learning attitudes, and course satisfaction; qualitative data were collected through focus group interviews to gain a deeper understanding of students' learning experiences and course suggestions.
  Interventions: Behavioral: Geriatric Ｂeauty and Ｈealth Care Learning Program

INTERVENTIONS:
Behavioral: Geriatric Ｂeauty and Ｈealth Care Learning Program — An educational course on geriatric care designed to enhance students' attitudes toward older adults and learning outcomes. The intervention includes lectures, group discussions, and interactive learning activities. Effectiveness is measured using pre- and post-course surveys and focus group interviews.

SUMMARY:
This study develops and evaluates a "Senior Beauty and Health Care" course designed to improve students' awareness, attitudes, and skills in caring for older adults' appearance and well-being. Using experiential learning and community practice, the course aims to reduce negative stereotypes and boost students' motivation and competence. A mixed-methods approach, including pretest-posttest surveys and focus group interviews, will assess the course's effectiveness and provide insights for future geriatric care education.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old. Conscious and able to communicate in Mandarin or Taiwanese. Provided informed consent after being informed of the study purpose.

Exclusion Criteria:

* Refusal to provide consent or students currently on leave of absence will not be enrolled.

Diagnosed by a physician with severe mental illness or otherwise deemed unsuitable for participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 65 (Estimated)
Dates: Start 2025-09-18 (Estimated); Primary Completion 2026-01-23 (Estimated); Study Completion 2026-01-23 (Estimated)

PRIMARY OUTCOMES:
Change in students' attitudes toward older adults | At baseline (pre-course) and immediately after course completion
  Measured using a validated attitude scale assessing stereotypes and perceptions of older adults before and after the course intervention.
Change in students' learning attitudes and motivation | At baseline and immediately post-course.
  Assessed via a standardized questionnaire measuring learning motivation, engagement, and confidence before and after the intervention.

SECONDARY OUTCOMES:
Qualitative feedback on learning experiences and course design | Within 2 weeks after course completion.
  Explored through focus group interviews to gather in-depth perceptions, reflections, and suggestions for course improvement.

CONTACTS AND LOCATIONS:
Locations (1):
- Chang Gung University of Science and Technology, Taoyuan District, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided